CLINICAL TRIAL: NCT05525767
Title: Prospective, Multicenter, Single-arm Clinical Study of Chemotherapy Combined With Bevacizumab Neoadjuvant Therapy for Early or Locally Advanced HER2-negative Breast Cancer
Brief Title: Chemotherapy Combined With Bevacizumab Neoadjuvant Therapy for HER2-negative Breast Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021198-1
Record Dates: First submitted 2022-08-28; First posted 2022-09-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): Bevacizumab 10mg/Kg d1, 1/21d
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — All subjects enrolled will receive bevacizumab .Subjects continued to take medication until disease progression, unacceptable toxicity, withdrawal of informed consent, or discontinuation of medication at the discretion of the investigator.

SUMMARY:
This is an prospective, multicenter, single-arm clinical study.

DETAILED DESCRIPTION:
Prospective, multicenter, single-arm clinical study of chemotherapy combined with bevacizumab neoadjuvant therapy for early or locally advanced HER2-negative breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Signed the informed consent and volunteered to join the study with good compliance;

3, histopathologically confirmed HER2-negative invasive breast cancer (including triple-negative breast cancer; Or Luminal breast cancer, that is, ER/PR positive and HER2 negative) :

* HER2 negative was defined as 0/1+ on standard IHC test; HER2/CEP17 ratio was less than 2.0 or HER2 gene copy number was less than 4.
* ER positive and/or PR positive were defined as the proportion of positively stained tumor cells in all tumor cells ≥1%;

  4. According to the American Joint Committee on Cancer (AJCC) 8th edition TNM stage II-IIIC (T2-T4 plus any N, or any T plus N1-3, M0);

  5. The main organs function well and meet the following standards:

A) Hemoglobin (HGB)≥90g/L;

B) Neutrophil absolute value (NEUT)≥1.5×109/L;

C) Platelet count (PLT)≥ 100×109/L;

D) leukocyte ≥3.0×109/L;

E) Total bilirubin <1.5 ULN (upper limit of normal)

F) Creatinine < 1.5×ULN

G) AST/ALT < 1.5×ULN;

6. Cardiac ultrasound: left ventricular ejection fraction (LVEF≥55%);

7. The investigators determined that the patients were suitable for treatment with bevacizumab.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer;
2. Received treatment for the disease, including chemotherapy, endocrine therapy, radiotherapy, immunotherapy, etc.;
3. Patients who are participating in other intervention studies;
4. Women with confirmed pregnancy or lactation;
5. According to the judgment of the investigator, the subjects have concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or the subjects think that there are other reasons that are not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PCR | 24 months
  pathologic complete response

SECONDARY OUTCOMES:
ORR | 24 months
  objective response rate
AE Advese Event Advese Event breast conservation rates | 24 months
  Advese Event
BCR breast conservation rates | 24 months
  breast conservation rates

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No